CLINICAL TRIAL: NCT00113685
Title: Effect of Hypertonic Resuscitation for Blunt Trauma
Brief Title: Hypertonic Saline With Dextran for Treating Hypovolemic Shock and Severe Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eileen Bulger, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20737; R01HL073233 (NIH)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Head Injuries, Closed; Shock; Shock, Traumatic
MeSH Terms: conditions — Respiratory Distress Syndrome; Head Injuries, Closed; Shock; Shock, Traumatic | interventions — hypertonic saline-dextran solution; Ringer's Lactate

INTERVENTIONS:
Drug: Hypertonic Saline-Dextran Solution
Drug: Lactated Ringer's Solution

SUMMARY:
The purpose of this study is to evaluate the clinical outcome of patients following blunt traumatic injury with hypovolemic shock, who receive either lactated ringer's solution or hypertonic saline with dextran (HSD) resuscitation; also, to focus specifically on neurologic outcome in patients with brain injury and on the effect of HSD resuscitation on inflammatory cell responsiveness.

DETAILED DESCRIPTION:
BACKGROUND:

Trauma is the leading cause of death among Americans between the ages of 1 and 35 years. The majority of these deaths result from hypovolemic shock, a type of shock in which the heart is unable to supply enough blood to the body, and the resulting severe brain injury. Patients in hypovolemic shock develop a state of systemic tissue ischemia with a subsequent reperfusion injury at the time of fluid resuscitation. Conventional resuscitation of these patients involves the intravenous administration of a large volume of isotonic or slightly hypotonic (lactated ringers) solutions beginning in the pre-hospital environment. Previous studies have suggested that an alternative resuscitation fluid, HSD, may reduce mortality in these patients; but these studies have not been conclusive. Furthermore, HSD may have specific advantages in the brain-injured patient, as it may aid in the rapid restoration of cerebral perfusion, prevent extravascular fluid sequestration, and thus, limit secondary brain injury. In addition, recent studies have demonstrated that hypertonicity significantly alters the activation of inflammatory cells, which may result in a reduction in subsequent organ injury following whole body ischemia/reperfusion and ultimately decrease nosocomial infection rates.

Blunt trauma victims with low blood pressures will be identified by pre-hospital providers (paramedics and flight nurses) and randomized to receive either 250 cc of HSD or 250 cc of isotonic solution (lactated ringer's solution). Lactated ringer's solution is the current standard of care with which the ambulances and helicopters will be supplied. All bags of study solution will be prepared by the Harborview Medical Center pharmacy.

DESIGN NARRATIVE:

This randomized clinical trial seeks to evaluate the clinical outcome and inflammatory cell function of patients in shock following blunt traumatic injury who are randomized to receive either 7.5% hypertonic saline/6% dextran (HSD) followed by lactated ringer's solution or lactated ringer's solution alone. It is hypothesized that HSD resuscitation will inhibit the initial excessive systemic activation of the inflammatory response, which will translate into a reduction in the incidence of organ dysfunction typically induced by this response. Furthermore, the study will evaluate the impact of HSD resuscitation on recovery following traumatic brain injury, as previous studies suggest that this subgroup has the greatest survival advantage from HSD intervention. The specific aims for this study include the following: Aim 1: To determine the impact of pre-hospital administration of HSD on the development of organ failure following blunt traumatic injury with hypovolemic shock. Aim 2: To determine the impact of pre-hospital administration of HSD on the neurologic outcome following brain injury for patients in hypovolemic shock. Aim 3a: To determine the effect of pre-hospital administration of HSD on the activation of circulating neutrophils and monocytes. Aim 3b: To determine the effect of pre-hospital administration of HSD on the activation of T lymphocytes. The study builds upon previous research that has demonstrated the safety and practicality of this resuscitation strategy in the pre-hospital environment. A more detailed understanding of the immuno-inflammatory effects of hypertonicity for all patients and the long-term neurologic outcome for patients with brain injury is critical for determining the role of this resuscitation approach in such critically injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Recent blunt trauma
* Of adult size if age is unknown
* Pre-hospital systolic bloood pressure 90 mm Hg or less
* Altered mental status
* Transported directly to Harborview Medical Center from the injury event

Exclusion Criteria:

* Ongoing CPR
* Transferred from outside hospitals
* Pregnant or suspected pregnancy
* Presence of injuries from penetrating trauma
* Receiving more than 2000 cc of crystaloid prior to study fluid administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209
Dates: Start 2003-04; Study Completion 2007-03

PRIMARY OUTCOMES:
Adult respiratory distress syndrome symptoms (measured 28 days post-injury)

SECONDARY OUTCOMES:
Multiple organ failure syndrome
28 day mortality
Nosocomial infections
Duration of hospital and ICU stay
Duration of mechanical ventilation
Neurologic outcome for patients with traumatic brain injury based on the Glasgow Outcome Score and Disability Rating Score (measured at 6 and 12 months post-injury)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Bulger, Study Chair — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Bulger EM, Jurkovich GJ, Nathens AB, Copass MK, Hanson S, Cooper C, Liu PY, Neff M, Awan AB, Warner K, Maier RV. Hypertonic resuscitation of hypovolemic shock after blunt trauma: a randomized controlled trial. Arch Surg. 2008 Feb;143(2):139-48; discussion 149. doi: 10.1001/archsurg.2007.41. PMID 18283138